CLINICAL TRIAL: NCT05616572
Title: Online Educational Tool to Increase Knowledge and Decrease Anxiety in Caregivers of Pediatric Oncology Patients
Brief Title: Online Educational Tool for Caregivers of Pediatric Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202207059
Record Dates: First submitted 2022-11-02; First posted 2022-11-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Caregiver Burden; Care Giving Burden; Pediatric Cancer
Keywords: caregiver; pediatric oncology
MeSH Terms: conditions — Caregiver Burden; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregiver (Experimental): After consent, the study visit will occur. The study visit will consist of a brief set of demographic questions and a pre-game play knowledge assessment and anxiety assessment, followed by completion of the OncoWhiz game. Immediately after utilizing OncoWhiz, the participant will complete a knowledge assessment and anxiety assessment, in addition to a satisfaction survey.
  Interventions: Behavioral: OncoWhiz

INTERVENTIONS:
Behavioral: OncoWhiz — OncoWhiz is an online educational tool designed to supplement current institutional caregiver education. OncoWhiz requires low graphical demands, has no-end user downloads, and is compatible with both desktop and mobile phones. Questions are derived from the institutional binder and are written at a fifth-grade reading level for user accessibility.

SUMMARY:
The goal of this study is to assess the feasibility of using a game-based tool for caregivers of pediatric oncology patients to increase caregiver knowledge about supportive care for oncology patients while simultaneously reducing caregiver anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of a pediatric cancer patient who was recently diagnosed with cancer, including all pediatric malignancies. Multiple caregivers can be enrolled. Caregiver is defined as a person who is responsible for the direct care, protection, and supervision of the pediatric cancer patient. In this context, a caregiver is not required to be the parent or legal guardian.
* Caregivers must have completed oncology nursing education either in the inpatient or outpatient setting.

  * Inpatient setting: Before discharge from hospital after nursing education
  * Outpatient setting: Within 15 days of discharge from the inpatient setting after nursing education or within 21 days of nursing education if diagnosis made in the outpatient setting

Exclusion Criteria:

* If less than 18 years of age
* Unable to utilize the electronic tool, complete the pre/post questionnaires and anxiety scale due to reading abilities, intellectual or physical disabilities.
* Cared for another child with cancer or secondary diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of using game-based tool to augment oncological education in caregivers of children newly diagnosed with cancer as measured by percentage of caregivers that enroll and complete study visit. | Through completion of study visit (Day 1) for all participants (estimated to be 1 year)
Feasibility of using game-based tool to augment oncological education in caregivers of children newly diagnosed with cancer as measured by the average time to completion of the educational tool. | Through completion of study visit (Day 1) for all participants (estimated to be 1 year)
Feasibility of using game-based tool to augment oncological education in caregivers of children newly diagnosed with cancer as measured by average time to complete the study visit. | Through completion of study visit (Day 1) for all participants (estimated to be 1 year)

SECONDARY OUTCOMES:
Determine the impact of a game-based tool in decreasing anxiety of caregivers of children newly diagnosed with cancer as measured by change in anxiety. | Prior to OncoWhiz and after OncoWhiz (Day 1)
  Anxiety will be quantified by the State-Trait Anxiety Inventory (STAI) Form. Participants will answer 40 questions regarding how they generally feel. There are 2 subscales within this assessment, both consisting of 20 separate items on a 4-point scale. The State Anxiety Scale (Y-1) evaluates the current state of anxiety while the Trait Anxiety Scale (Y-2) evaluates anxiety-proneness as a personality trait. A higher score indicates greater anxiety.
Determine the impact of a game-based tool in increasing knowledge of caregivers of children newly diagnosed with cancer as measure by change in knowledge. | Prior to OncoWhiz and after OncoWhiz (Day 1)
  The knowledge assessment consists of 20 multiple choice questions related to caregiving for children with cancer. The percentage of questions answered correctly before and after utilization of the tool will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Fields, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlies the published results will be available after deidentification.
Time Frame: The shared data will be available 6 months after publication, ending 36 months after article publication.
Access Criteria: These data will be available to researchers that provide a methodologically sound proposal. The data will be available to achieve the aims of the approved proposal. Proposals should be directed to fields_m@wustl.edu.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu